CLINICAL TRIAL: NCT02962453
Title: Multi-Modalities Evaluation of Gait Rehabilitation Robot of an End-Effector on Neuro-Muscular Pathway of the Proximal Muscles in Patients After Total Knee Arthroplasty
Brief Title: Evaluation of Gait Rehabilitation Robot of an End-Effector on Neuro-Muscular Pathway in Patients After Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Chang Ho Hwang, Associated Professor, Ulsan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: chhwang6
Record Dates: First submitted 2016-11-02; First posted 2016-11-11 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morning walk (Experimental): Rehabilitation using end-effector type gait robot for 5days.
  Interventions: Device: Morning walk
- Ground Walker (Active Comparator): Rehabilitation using walker for 5days.
  Interventions: Device: Ground Walker

INTERVENTIONS:
Device: Morning walk — gait training with Morning walk three times during 5 minutes with 5 minute break a day over 5 weekdays
  Other Names: end-effector type robot
  Arms: Morning walk
Device: Ground Walker — gait training with ground walker until corresponding 200 steps during 5 minutes with 5 minute break a day over 5 weekdays
  Arms: Ground Walker

SUMMARY:
The aim of this study is to determine the clinical efficacy of gait rehabilitation robot through cortico-spinal-muscular pathway activation of the muscles remotely located from the end-effecter in patients after total knee arthroplasty.

DETAILED DESCRIPTION:
pre-interventional evaluation; within 1 day of intervention start primary end point; 3 days after intervention start secondary end point; 5 days after intervention start

ELIGIBILITY:
Inclusion Criteria:

* Patients after Unilateral Total Knee Arthroplasty

Exclusion Criteria:

* brain disease, spinal cord injury, peripheral neuropathy, myopathy
* Inability to ambulate fully due to muscukoskeletal disorders
* MMSE<23
* history of arthroplasty surgery on either of legs
* Cardiac pacemaker
* Refusal of participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11; Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Change of Isometric muscle strength | 0 day( within 6 hours before the treatment start) and 5 day(within 6 hours after treatment stop)
  peak torque (Nm/㎡), Maximal ratio of torque development (RTD) (degree/sec)

SECONDARY OUTCOMES:
Change of Cortico-motor Excitability | 0 day( within 6 hours before the treatment start) and 5 day(within 6 hours after treatment stop)
  maximum & mean amplitude of peak to peak MEP (mV and mV), amplitude of peak to peak MEP/maximum M-wave (mV/mV)
Change of Spinal Motor-neuron Excitability | 0 day( within 6 hours before the treatment start) and 5 day(within 6 hours after treatment stop)
  Peak to peak Max. H-reflex (mV/mV), Peak to peak Max. H-wave/Max. M-reflex (mV/mV*㎡)
Change of Cross-sectional area and volume of thigh muscle | 0 day( within 6 hours before the treatment start) and 5 day(within 6 hours after treatment stop)
  Cross-sectional area (c㎡) and and volume (cm3)
Change of Muscle work | 0 day( within 6 hours before the treatment start) and 5 day(within 6 hours after treatment stop)
  peak and mean amplitude of CMAP (mV and mV) and mean area & total area of CMAP (c㎡/sec and c㎡/sec)

CONTACTS AND LOCATIONS:
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea

IPD SHARING:
Plan to Share IPD: No